CLINICAL TRIAL: NCT04580095
Title: Technology Revisiting Ultrasound Solutions of Tomorrow - Artificial Intelligence for Improved Echocardiography
Brief Title: Artificial Intelligence for Improved Echocardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TRUST-AI_201
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With AI algorithm (Experimental): In the "With AI algorithm" arm, the sonographer will perform the echocardiographic exam using the AI algorithm.
  Interventions: Other: AI algorithm for apical foreshortening in echocardiography
- Without AI algorithm (No Intervention): In the "Without AI algorithm", the echocardiographic exam will be performed without the use of the AI algorithm.

INTERVENTIONS:
Other: AI algorithm for apical foreshortening in echocardiography — The algorithm is based on artificial intelligence, giving the sonographer performing the echocardiographic exam real-time feedback on left ventricular apical foreshortening.The algorithm is developed using deep learning techniques by technologists at the Department of Circulation and Medical Imaging, NTNU.
  Arms: With AI algorithm

SUMMARY:
The purpose of this study is to assess the effect of artificial intelligence algorithms on image quality in echocardiography.

DETAILED DESCRIPTION:
The study population will be recruited from appointed patients at the Clinic of Cardiology, St. Olavs Hospital. After being informed about the study, all patients giving informed consent and meeting the eligibility requirements will undergo their standard clinical echocardiographic exam performed by a sonographer at the clinic. Two additional examinations will then be performed by a different sonographer and an expert cardiologist, respectively.

In one of the study arms the sonographer randomized to perform the second exam will use the AI algorithm (intervention).

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent

Exclusion Criteria:

* Indication for echocardiographic contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Left ventricular apical foreshortening | 0 days
  Apical foreshortening will be evaluated in a blinded manner by echocardiography experts post hoc. The two study arms will be compared.

OTHER OUTCOMES:
Image quality | 0 days
  Image quality will be evaluated in a blinded manner by echocardiography experts post hoc. A standardized scoring system for image quality in echocardiography developed locally will be utilized for evaluation with score 1-6, where 1 is minimum and 6 is maximum score. The two study arms will be compared.
Inter-observer variation of left ventricular size | 0 days
  Throughout this study, the sonographers and expert cardiologist will perform measurements based on their individual echocardiographic images. Differences in measurements will be evaluated to determine inter-observer variation between sonographers and cardiologists.
Inter-observer variation of left ventricular function | 0 days
  Throughout this study, the sonographers and expert cardiologist will perform measurements based on their individual echocardiographic images. Differences in measurements will be evaluated to determine inter-observer variation between sonographers and cardiologists.
Validation of AI algorithm to detect foreshortening | 0 days
  Comparison of AI algorithm to detect foreshortening with manual reference
Inter-observer variation of left atrial size | 0 days
  Throughout this study, the sonographers and expert cardiologist will perform measurements based on their individual echocardiographic images. Differences in measurements will be evaluated to determine inter-observer variation between sonographers and cardiologists.
Inter-observer variation of left atrial function | 0 days
  Throughout this study, the sonographers and expert cardiologist will perform measurements based on their individual echocardiographic images. Differences in measurements will be evaluated to determine inter-observer variation between sonographers and cardiologists.
Development of AI algorithm for real-time assessment of left atrium | 0 days
  Cardiac structures as left atrial (LA) lumen, LA wall, LA appendix, mitral valve will be annotated and used as reference.
Variation by methodology | 0 days
  Variation in measurement by the mode of measurement

CONTACTS AND LOCATIONS:
Locations (1):
- St. Olav University Hospital, Trondheim, Norway

REFERENCES:
- [Derived] Pettersen H, Sabo S, Pasdeloup D, Smistad E, Olaisen S, Ostvik A, Stolen S, Grenne BL, Lovstakken L, Dalen H, Holte E. Real-time deep learning-based image guiding and automated left ventricular measurements to reduce test-retest variability. Open Heart. 2025 Dec 7;12(2):e003783. doi: 10.1136/openhrt-2025-003783. PMID 41360622
- [Derived] Sabo S, Pasdeloup D, Pettersen HN, Smistad E, Ostvik A, Olaisen SH, Stolen SB, Grenne BL, Holte E, Lovstakken L, Dalen H. Real-time guidance by deep learning of experienced operators to improve the standardization of echocardiographic acquisitions. Eur Heart J Imaging Methods Pract. 2023 Nov 27;1(2):qyad040. doi: 10.1093/ehjimp/qyad040. eCollection 2023 Sep. PMID 39045079
- [Derived] Sabo S, Pettersen HN, Smistad E, Pasdeloup D, Stolen SB, Grenne BL, Lovstakken L, Holte E, Dalen H. Real-time guiding by deep learning during echocardiography to reduce left ventricular foreshortening and measurement variability. Eur Heart J Imaging Methods Pract. 2023 Aug 1;1(1):qyad012. doi: 10.1093/ehjimp/qyad012. eCollection 2023 May. PMID 39044792